CLINICAL TRIAL: NCT03652129
Title: Digitized Assessment for the Survival of Mature Anterior Teeth With Periapical Lesion After One Step Regenerative Approach Using Different Asepsis Maneuvers
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Mohsen Abielhassan, Assisstant Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Regerative Endodontics
Record Dates: First submitted 2018-08-28; First posted 2018-08-29 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Dental Pulp Necrosis; Dental Pulp Disease; Dental Pulp; Degeneration
MeSH Terms: conditions — Dental Pulp Necrosis; Dental Pulp Diseases | interventions — Disinfection

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Laser Group (Experimental): Disinfection using biostimulating LASER
  Interventions: Procedure: Disinfection
- Nano irrigant Group (Experimental): Disinfection using Nano irrigant
  Interventions: Procedure: Disinfection
- Conventional irrigation protocol group (Active Comparator): disinfection using normal irrigation protocols
  Interventions: Procedure: Disinfection

INTERVENTIONS:
Procedure: Disinfection — Disinfection maneuver using LASER and nano irrigant

SUMMARY:
Trial is designed to allow revascularization and tissue engineering in necrotic teeth with peripical lesion in a single visit approach. different disinfection protocols is used to ensure that adequate disinfection of root canals is achieved to allow stem cells to differentiate and proliferate generating pulp like tissue and turning back tooth to live with periapical healing of resorbed bone.

DETAILED DESCRIPTION:
Preservation of the natural dentition had always been a primary objective in endodontic practice. When the pulp is diseased or requires removal for restorative reasons, it is replaced with an artificial filling material during conventional root canal treatment. Root canal treatment has lots of controversies, starting with weakening of remaining tooth structure, affecting the tooth survival. Also Root canal treated teeth are considered to be weaker than vital tooth, requiring the placement of a post and core, which itself is doubtful whether it increases fracture resistance of the tooth or it weakens it.1 The most important controversy is that the survival of affected pulp is hindered by the conventional root canal treatment2. Thus a new treatment approach was introduced utilizing the body ability to regenerate, called Pulp Regeneration. Regeneration was first introduced in the dental field as a solution for immature apex treatment, as it is very difficult to treat them using the conventional root canal treatment3 American Dental Association adopted the tissue engineering concept and pulp regeneration in 20114. Regeneration was focused on the treatment of immature necrotic teeth so as to allow root completion, improving both the functionality and durability of the affected tooth. Depending on the success of pulp regeneration in treating immature teeth, ambitious dentists started to look forward on treating mature teeth as a substitution to the conventional root canal treatment. 5

A shift to tissue engineering took place. Utilizing a blood clot in the affected tooth with immature roots was very beneficial, as it acts as a scaffold for the migration of stem cells and morphogens to allow regeneration .6 On the other hand, lots of clinicians were very doubtful about treating mature teeth with the same protocol, as the small apical foramen might not provide a good portal for the entry of stem cells and growth factors, which in turn is very important for the success of pulp regeneration.7

These doubts encouraged researchers to look for an alternative to the stem cells other than the apical papilla, from this concept the idea for using an alternative source of stem cells and growth factors as platelet rich plasma (PRP) emerged. The use of Platelet Rich Plasma (PRP) as a potentially ideal scaffold for regenerative endodontic therapy has been documented8. However, the use of bovine thrombin for the activation of PRP has been an issue of controversy, as it requires non autologous anticoagulant known to hinder the process of pulp regeneration 9.

This led to the development of the second generation, Platelet concentrate known as Choukroun's Platelet Rich Fibrin (PRF) which is totally autologous in nature. Platelet rich fibrin (PRF) was very promising, but it is debatable whether to use PRP or PRF10. One protocol of the regenerative approach is the use of Antibiotic paste as intra canal medicament in a 2 step procedures, due to the world wide trend of limitation of the use of antibiotics systemically and locally the assessment of the outcome of single visit regenerative approach is mandatory, and because the main limitation for such intervention is adequate disinfection of root canal assessment of different asepsis maneuvers is also of great importance since literature and evidence based information lack any studies assessing such techniques.

The clinician at the end of this study must determine which disinfection protocol allows for more survival of tooth, revitalization of the affected mature tooth and faster healing of periapical lesion following one step regenerative approach. Healing will be measured using digital radiography and cone beam computed topography11. Repair of the tooth neural innervation will be tested by electric pulp tester12.

ELIGIBILITY:
Inclusion criteria:

* Patients who are free from any physical or mental handicapping condition with no underlying systemic diseases.
* Non-pregnant females
* Single canalled anterior teeth.
* Patients having non-vital, mature, anterior teeth, radiographic evidence of periapical lesion.
* Positive patient/Guardian compliance for participation in the study.

Exclusion criteria:

* Any known sensitivity or adverse reactions to medicaments or pharmaceuticals necessary to complete the trial.
* Non-restorable coronal portion of teeth involved in the trial.
* Vital teeth
* immature teeth
* Traumatized teeth
* Radiographic evidence of external or internal root resorption.
* Any criterion, not mentioned in the inclusion criteria

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2018-08-22 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Periapical Healing | 1 year
  Bone healing

SECONDARY OUTCOMES:
Survival of tooth | 1 year
  tooth survival after procedure
Sensitivity | 1 year
  assess sensitivity using pulp tester

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided